CLINICAL TRIAL: NCT04001582
Title: The UK Facioscapulohumeral Muscular Dystrophy Patient Registry
Brief Title: The United Kingdom Facioscapulohumeral Muscular Dystrophy Patient Registry
Status: Recruiting | Type: Observational
Sponsor: Newcastle University (Other)
Responsible Party: Sponsor
Other Study IDs: 18/NE/0288
Record Dates: First submitted 2019-06-25; First posted 2019-06-28 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Facioscapulohumeral Muscular Dystrophy
Keywords: FSHD; Facioscapulohumeral Muscular Dystrophy; Facioscapulohumeral Muscular Dystrophy Type 1; Facioscapulohumeral Muscular Dystrophy Type 2; Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Facioscapulohumeral; Muscular Dystrophies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 99 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with FSHD: Patients with a confirmed or pending diagnosis of FSHD, living in the UK are eligible to join the registry. Parents/guardians can register a child under 16 years old.
  Interventions: Other: Patient Registry

INTERVENTIONS:
Other: Patient Registry — Participants who have volunteered to participate will complete various questionnaires relating to their condition.

SUMMARY:
Facioscapulohumeral Dystrophy (FSHD) is the third most common form of neuromuscular dystrophy worldwide with an estimated prevalence of one in 20,000. FSHD is an autosomal dominant genetic disease and is estimated to affect up to 3,000 people in the UK.

The patient registry facilitates a questionnaire based research study to better characterise and understand the disease in the UK, and helps to identify potential participants eligible for clinical trials.

DETAILED DESCRIPTION:
The UK FSHD Patient Registry (https://www.fshd-registry.org/uk/) recruits any individual, from anywhere within the United Kingdom, with a diagnosis of FSHD. The registry is sponsored by Muscular Dystrophy UK. Participants may be referred to the registry by health care professionals, genetic testing/laboratory centres who are aware of the registry etc. Alternatively, a participant may have discovered the registry via promotional activities or by their own online searches. After completing the consent process, participants are able to enter information on to the registry platform (note all forms are available to view on the registry website before joining the registry). This is an ongoing database and all participants are invited to update their information on an annual basis.

The database is designed to be self reporting, however where specialised clinical or genetic information is required, the neuromuscular specialist in charge of the participants care can be invited to provide some additional information. The participant is able to select a health care provider from a pre-populated list at registration stage, if they wish to (optional feature). This information is included in the patient information and consent. Relevant R&D approval has been recieved.

ELIGIBILITY:
Inclusion Criteria:

- All patients with a confirmed FSHD diagnosis (or pending diagnosis) who reside in the UK are eligible for inclusion.

Exclusion Criteria:

* Any confirmed NMD other than FSHD
* Living outside of the UK

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with FSHD volunteer to participate in this study. The registry is advertised through neuromuscular disease clinics, the registry website, patient organisations and conferences and meetings throughout the UK.
Sampling Method: Non-Probability Sample
Enrollment: 1018 (Estimated)
Dates: Start 2013-05 (Actual); Primary Completion 2040-01 (Estimated); Study Completion 2040-01 (Estimated)

PRIMARY OUTCOMES:
Patient questionnaire | 12 months
  Patient reported FSHD clinical diagnosis, symptoms relating to muscle weakness, motor function, ventilation, retinal vascular disease, hearing loss, scapular fixation, family history and ethnicity.
McGill Pain Questionnaire | 12 months
  Patient reported current pain.
FSHD Pain Questionnaire | 12 months
  Patient reported experience of pain.
The Short Form Health Survey (SF-36) | 12 months
  Patient reported quality of life.
The Individualized Neuromuscular Quality of Life questionnaire (INQoL) | 12 months
  Patient reported quality of life.
Scapular fixation questionnaire | 12 months
  Patient reported experience of scapular fixation surgery.
Clinician questionnaire | 12 months
  Clinician reported genetic confirmation of FSHD.

CONTACTS AND LOCATIONS:
Overall Officials: Chiara Marini-Bettolo, MD, PhD, Principal Investigator — John Walton Muscular Dystrophy Research Centre
Locations (1):
- John Walton Muscular Dystrophy Research Centre, Newcastle upon Tyne, United Kingdom

REFERENCES:
- [Result] Moris G, Wood L, FernaNdez-Torron R, Gonzalez Coraspe JA, Turner C, Hilton-Jones D, Norwood F, Willis T, Parton M, Rogers M, Hammans S, Roberts M, Househam E, Williams M, Lochmuller H, Evangelista T. Chronic pain has a strong impact on quality of life in facioscapulohumeral muscular dystrophy. Muscle Nerve. 2018 Mar;57(3):380-387. doi: 10.1002/mus.25991. Epub 2017 Nov 7. PMID 29053898
- [Result] Ricci G, Cammish P, Siciliano G, Tupler R, Lochmuller H, Evangelista T. Phenotype may predict the clinical course of facioscapolohumeral muscular dystrophy. Muscle Nerve. 2019 Jun;59(6):711-713. doi: 10.1002/mus.26474. Epub 2019 Apr 4. PMID 30895627
- [Result] Evangelista T, Wood L, Fernandez-Torron R, Williams M, Smith D, Lunt P, Hudson J, Norwood F, Orrell R, Willis T, Hilton-Jones D, Rafferty K, Guglieri M, Lochmuller H. Design, set-up and utility of the UK facioscapulohumeral muscular dystrophy patient registry. J Neurol. 2016 Jul;263(7):1401-8. doi: 10.1007/s00415-016-8132-1. Epub 2016 May 9. PMID 27159994
- See also: The UK FSHD Patient Registry website — https://www.fshd-registry.org/uk/